CLINICAL TRIAL: NCT06527508
Title: Construct Validity and Intra-Observer Reliability of the Self-Report Version of Strengths and Difficulties Questionnaire in Children With Cerebral Palsy
Brief Title: Construct Validity and Intra-Observer Reliability of the SDQ
Status: Completed | Type: Observational
Sponsor: Bingol University (Other)
Responsible Party: Principal Investigator, Hasan Bingöl, Assistant Professor, Bingol University
Other Study IDs: E-33117789-044-167349
Record Dates: First submitted 2024-07-25; First posted 2024-07-30 (Actual); Last update posted 2024-07-30 (Actual); Status verified 2024-07

CONDITIONS: Cerebral Palsy
Keywords: cerebral palsy; Strength and Difficulties Questionnaire; validity; reliability
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Non-Interventional — This study has a observational design

SUMMARY:
The aim of the observational study is to investigate the validity and reliability of a self-report version of the Strength and Difficulties Questionnaire (SDQ) for 11-17 years in children with cerebral palsy (CP). That is, the current study explore if the self-report version of the SDQ would be valid and reliable in children with CP to report their mental health problems themself

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of CP, a communication level of I-III on the Communication Function Classification System (CFCS), and no severe intellectual disability

Exclusion Criteria:

* the presence of an inability to comprehend items on the SDQ and involuntary attendance of a possible re-test after two weeks (i.e., for re-test reliability)

Ages: 11 Years to 17 Years | Sex: All
Age Groups: Child
Study Population: The study included children aged 11-17 years who were diagnosed with CP by health science boards at the government or education and research hospitals.
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-05-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Change from baseline in mental health on the 3-point Strength and Difficulties Questionnaire (SDQ) at 2 week | Baseline and Week 2
  The Strength and Difficulties Questionnaire (SDQ) was created by Goodman as a brief screening tool for assessing emotional and behavioral problems in children and adolescents. There are two primary versions of the SDQ, self-report and proxy-report, for different age bands: 2-4, 11-17, 4-17 and over 18 years. The SDQ consists of subscales for emotional problems, conduct problems, hyperactivity-inattention problems, peer problems, and prosocial scales. Each subscale comprises five items, with 'somewhat true' being always scored as 1. On the other hand, the scoring for 'not true' and 'certainly true' varied depending on the item (i.e., 0 or 2).

CONTACTS AND LOCATIONS:
Locations (1):
- Bingöl University, Bingöl, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Downs J, Blackmore AM, Epstein A, Skoss R, Langdon K, Jacoby P, Whitehouse AJO, Leonard H, Rowe PW, Glasson EJ; Cerebral Palsy Mental Health Group. The prevalence of mental health disorders and symptoms in children and adolescents with cerebral palsy: a systematic review and meta-analysis. Dev Med Child Neurol. 2018 Jan;60(1):30-38. doi: 10.1111/dmcn.13555. Epub 2017 Sep 15. PMID 28914445
- [Result] Anthoine E, Moret L, Regnault A, Sebille V, Hardouin JB. Sample size used to validate a scale: a review of publications on newly-developed patient reported outcomes measures. Health Qual Life Outcomes. 2014 Dec 9;12:176. doi: 10.1186/s12955-014-0176-2. PMID 25492701
- [Derived] Bingol H, Karaoba DD. Reliability and Construct Validity of the Self-Report Version of Strengths and Difficulties Questionnaire in Children and Adolescents With Cerebral Palsy. Child Care Health Dev. 2025 Jul;51(4):e70114. doi: 10.1111/cch.70114. PMID 40490683